CLINICAL TRIAL: NCT01546311
Title: Evaluation of a Pro-Active Dynamic Accommodating Socket
Acronym: PADS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Infoscitex Corporation (Industry)
Collaborators: Liberating Technologies, Inc. (Industry); Telemedicine & Advanced Technology Research Center (Other)
Responsible Party: Principal Investigator, Kristen Leroy, Group Leader, Biomedical Devices, Infoscitex Corporation
Other Study IDs: IST1387 PADSII; W81XWH-09-C-0028 (Other Grant/Funding Number: US Army MRMC)
Record Dates: First submitted 2012-03-02; First posted 2012-03-07 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Amputation
Keywords: prosthetic socket; residual limb volume fluctuation; instantaneous bladder

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- lower limb amputees
  Interventions: Device: Pro Active Dynamic Accommodating Socket

INTERVENTIONS:
Device: Pro Active Dynamic Accommodating Socket — Socket with bladders that instantaneously adjusts to volume fluctuations in the residual limb

SUMMARY:
The primary objective of this study is to assess the effectiveness of the pro-active dynamic socket (PADS) on increasing socket comfort and fit for transfemoral and transtibial amputees during ambulation and rest, addressing residual limb volume fluctuations with a controlled flow bladder system.

DETAILED DESCRIPTION:
The purpose of this study is to compare a pro-active dynamic socket to each user's everyday ischial containment socket in above-knee amputees, or transtibial socket in below-knee amputees. It is the goal for the pro-active dynamic socket to alleviate high pressure on the residual limb and improve socket fit and comfort. The pro-active dynamic socket contains bladders that can inflate and deflate throughout the gait cycle to appropriate levels of pressure to improve socket fit. These improvements will be confirmed by pressure measurements on the distal end of the residual limb, the ischium, and the bladders located around the socket walls.

ELIGIBILITY:
Inclusion Criteria:

* transfemoral or transtibial amputation
* unilateral or bilateral amputation
* stable residual limb volume
* read, write, and speak English for proper consent and responding to questionnaire

Exclusion Criteria:

* evidence or history of residual limb skin conditions such as irritation or sores
* presence of phantom limb pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Persons with transfemoral or transtibial amputation who have been using a prosthesis for at least one month will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Estimated)
Dates: Start 2012-01; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kristen J LeRoy, Principal Investigator — Infoscitex Corporation
Locations (2):
- United States (2):
  - Liberating Technologies, Inc, Holliston, Massachusetts
  - Next Step O&P, Newton, Massachusetts